CLINICAL TRIAL: NCT02322151
Title: Pharmacokinetics of Granulocyte Colony Stimulating Factor in the Breast Milk of Volunteer Peripheral Blood Stem Cell Donor
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 150047; 15-CC-0047
Record Dates: First submitted 2014-12-19; First posted 2014-12-23 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2016-10-14

CONDITIONS: Normal Physiology
Keywords: Filgrastim; Neupogen; Transplant; Breast Feeding; Concentration
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Background:

- The drug filgrastim (rGCSF) increases the number of blood-forming cells in the bloodstream. These cells can be collected from donors bloodstreams and used for transplant. Studies have shown that rGCSF is present in the breast milk of nursing mothers who are taking it. Based on these studies, it is now recommended that a nursing mother should not breastfeed from the time she receives the first dose of the drug until 2 days after the final dose. Researchers want to study the amount of the drug and its effect on the cells present in donor blood and breast milk. They hope to better understand the effects of this drug on breast milk.

Objectives:

- To understand the effects of filgrastim on breast milk.

Eligibility:

- Women enrolled in NIH protocol 00-CC-0165 and currently breastfeeding.

Design:

* Participants will receive rGCSF daily for 5 days. They will have blood taken daily.
* Participants will get a freezer bag containing 10 sterile, labeled containers for breast milk collection.
* Participants will transfer some of the breast milk they pump into one of the containers. They will write the date and time the milk was collected on the container. They will freeze the samples. Any remaining milk should be disposed of.
* Participants will bring the samples to NIH on the day of their stem cell collection procedure.
* For days 1 and 2 after stem cell collection, participants will continue to collect and freeze breast milk samples and dispose of any remaining milk.
* For days 3 5 after stem cell collection, participants will collect and freeze samples. They can also resume normal breastfeeding.
* A research nurse will arrange to collect the samples.

DETAILED DESCRIPTION:
Recombinant human granulocyte colony stimulating factor (rhGCSF) is routinely administered to volunteer peripheral blood stem cell (PBSC) donors in the National Marrow Donor Program (NMDP). Information about the excretion and pharmacokinetics of rhGCSF into human breast milk, however, is extremely limited. Two case reports exist, the first demonstrating only that subcutaneously administered rhGCSF is present in breast milk,1 and the second demonstrating that rhGCSF is not only present, but also remains in breast milk for two days after discontinuation of the medication.2 Based on the data from the latter case report, the NMDP suggests that donors abstain from breastfeeding during the administration of rhGCSF and for 48 hours after the last dose of rhGCSF is given. We intend to collect and test breast milk and peripheral blood from one volunteer NMDP donor during the course of her rhGCSF therapy and for 5 days thereafter, with the intention of better characterizing this rare and unique situation. Collected samples will be used for granulocyte colony stimulating factor (GCSF) quantitation and complete blood counts. Additionally, we will collect a single breast milk sample from three rhGCSF-na(SqrRoot) ve volunteers for use as negative control samples for assay calibration.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women enrolled in NIH protocol 00-CC-0165 and currently breastfeeding.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2014-12-12; Primary Completion 2015-11-09 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
Analysis of collected samples | Within one year

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Conry Cantilena, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Shibata H, Yamane T, Aoyama Y, Nakamae H, Hasegawa T, Sakamoto C, Terada Y, Koh G, Hino M. Excretion of granulocyte colony-stimulating factor into human breast milk. Acta Haematol. 2003;110(4):200-1. doi: 10.1159/000074226. No abstract available. PMID 14663166
- [Background] Kaida K, Ikegame K, Fujioka T, Taniguchi Y, Inoue T, Hasei H, Tamaki H, Yoshihara S, Kawase I, Ogawa H. Kinetics of granulocyte colony-stimulating factor in the human milk of a nursing donor receiving treatment for mobilization of the peripheral blood stem cells. Acta Haematol. 2007;118(3):176-7. doi: 10.1159/000109267. Epub 2007 Oct 3. No abstract available. PMID 17914246
- [Background] Pessach I, Shimoni A, Nagler A. Granulocyte-colony stimulating factor for hematopoietic stem cell donation from healthy female donors during pregnancy and lactation: what do we know? Hum Reprod Update. 2013 May-Jun;19(3):259-67. doi: 10.1093/humupd/dms053. Epub 2013 Jan 3. PMID 23287427